CLINICAL TRIAL: NCT00442897
Title: Evaluate The Lipid-Lowering Efficacy and Safety of Vytorin in Comparison With Atorvastatin in Hypercholesterolaemic Patients With Coronary Artery Disease
Brief Title: Vytorin (10/20 Or 10/40) Compared to Atorvastatin (10 mg or 20 mg) in Patients With Coronary Artery Disease (0653A-126)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-126; MK0653A-126; 2007_006
Record Dates: First submitted 2007-02-28; First posted 2007-03-05 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: simvastatin (+) ezetimibe
- 2 (Active Comparator)
  Interventions: Drug: Comparator: atorvastatin

INTERVENTIONS:
Drug: simvastatin (+) ezetimibe — simvastatin (+) ezetimibe 10/20mg, tablet, once daily, 12wks(sub group:24wks)
  Other Names: MK0653A; Vytorin®
  Arms: 1
Drug: Comparator: atorvastatin — atorvastatin 10mg, tablet, once daily, 12wks(sub group:24wks)
  Other Names: Lipitor®
  Arms: 2

SUMMARY:
Evaluate the proportion of hyperlipaemic persons with known coronary heart disease achieving ldl-c goal as defined by the national cholesterol education program (NCEP) adult treatment panel (ATP) III guidelines

ELIGIBILITY:
Inclusion Criteria:

* Patients who are naïve to lowering lipid agent
* Patients who are treated with lowering lipid agents and had a wash-out period for 4 weeks.

Exclusion Criteria:

* Impaired kidney function
* Increased liver enzyme levels
* Pregnant women
* Hypersensitivity to ezetimibe and other statin agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited between September 2006 and May 2008.
Pre-assignment Details: Patients who were naïve to lipid-lowering agent or patients who were treated with lipid-lowering agent and had 4 week' wash-out period were enrolled in the study. The eligible patients will be allocated to one of vytorin 10/20 or atorvastatin 10 mg group in 1:1 ratio.
Groups:
- Vytorin: Vytorin group- The eligible patients were allocated to one of vytorin 10/20 or atorvastatin 10 mg group in 1:1 ratio. If patients didn't achieve LDL-C < 100 mg/dl after 6 weeks of treatment, they received the double dosage of study drug for the next 6 weeks (vytorin 10/40 or atorvastatin 20 mg) and If patients achieved LDL-C < 100 mg/dl, they received the same dosage of study drug for the next 6 weeks. Patients who were allocated to vytorin had vytorin 10/20 mg or 10/40 mg tablet, orally, once a day.
- Atorvastatin: Atorvastatin group- Patients who were allocated to atorvastatin had atorvastatin 10 mg or 20 mg tablet, orally, once a day.
Period: Base Study (12 Week Follow-up)
Arm/Group | Vytorin | Atorvastatin
Started | 118 | 111
Completed | 101 | 99
Not Completed | 17 | 12
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 7 | 3
Not completed — Withdrawal by Subject | 9 | 8
Period: 24 Weeks Follow-up (3 Centers)
Arm/Group | Vytorin | Atorvastatin
Started | 35 (66 Patients did not continue in the additional 12 week extension, for the 24 weeks follow-up period.) | 34 (65 Patients did not continue in the additional 12 week extension, for the 24 weeks follow-up period.)
Completed | 29 | 28
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vytorin | Atorvastatin | Total
Number analyzed (Participants) | 118 | 111 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.89 (9.28) | 61.74 (9.94) | 61.30 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 53 | 110
  Male | 61 | 58 | 119
Baseline Low Density Lipoprotein-Cholesterol (LDL-C) allocation strata [Number; unit: Participants]
  LDL-C 130-159mg/dl | 64 | 61 | 125
  LDL-C 160-189mg/dl | 38 | 31 | 69
  LDL-C >=190mg/dl | 16 | 18 | 34
  LDL-C <130mg/dl | 0 | 1 | 1
Baseline values for Apolipoprotein B (Apo B) [Mean (Standard Deviation); unit: mg/dL] | 113.23 (30.97) | 110.63 (31.63) | 111.97 (31.25)
Baseline values for High-Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 48.23 (10.25) | 48.9 (13.01) | 48.55 (11.65)
Baseline values for LDL-C:HDL-C [Mean (Standard Deviation); unit: Ratio] | 3.54 (1.13) | 3.54 (1.04) | 3.54 (1.08)
Baseline values for Low-Density Lipoprotein Cholesterol(LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 164.11 (33.52) | 162.56 (26.75) | 163.36 (30.37)
Baseline values for Non HDL-C [Mean (Standard Deviation); unit: mg/dL] | 191.54 (38.25) | 190.72 (31.11) | 191.14 (34.88)
Baseline values for Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 241.4 (39.53) | 239.58 (30.86) | 240.51 (35.51)
Baseline values for Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 142 (86.27) | 144 (57.34) | 143 (73.69)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 24.97 (2.92) | 24.86 (2.64) | 24.92 (2.78)
Body Weight [Mean (Standard Deviation); unit: Kilograms (Kg)] | 64.61 (9.78) | 64.40 (10.51) | 64.51 (10.12)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 75.86 (10.16) | 77.74 (10.53) | 76.77 (15.98)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 126.44 (15.23) | 129.53 (16.65) | 127.94 (15.98)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reaching the LDL-C (Low Density Lipoprotein-Cholesterol) Goal (< 100 mg/dl) After 6 Weeks of Treatment
Description: Primary objective is to evaluate the proportion of patients achieving LDL-C target <100 mg/dl recommend in National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) after 6 weeks of treatment(vytorin 10/20 vs. atorvastatin 10 mg)
Time Frame: After 6 weeks of treatment
Population: The analysis used all patient treated (APT) approach which included all patients who had baseline measured right before randomization, have taken the study drug more than once after randomization and have one measurement after the initiation of the treatment.
Measure: Number; unit: Participants
Arm/Group | Vytorin | Atorvastatin
Number analyzed (Participants) | 107 | 101
Participants | 89 | 63
Statistical Analysis 1: Comparison: Vytorin vs Atorvastatin; Test type: Superiority or Other; Odds Ratio (OR) = 3.714, 95% CI [1.77 to 7.78] — Odds ratio was adjusted by baseline LDL strata

2. Secondary Outcome: Number of Participants Reaching the LDL-C Goal (< 100 mg/dl) After 12 Weeks of Treatment
Description: If patients didn't achieve LDL-C <100 mg/dl after 6 weeks of treatment, they received the double dosage of study drug for the next 6 weeks (vytorin 10/40 or atorvastatin 20 mg) and If achieved LDL-C < 100 mg/dl, they received the same dosage of study drug for the next 6 weeks.
Time Frame: After 12 weeks of the treatment
Population: All patient treated (APT) approach
Measure: Number; unit: Participants
Arm/Group | Vytorin | Atorvastatin
Number analyzed (Participants) | 107 | 101
Participants | 85 | 63
Statistical Analysis 1: Comparison: Vytorin vs Atorvastatin; Test type: Superiority or Other; Odds Ratio (OR) = 2.579, 95% CI [1.32 to 5.06] — Odds ratio was adjusted by baseline LDL strata

ADVERSE EVENTS:
Description: Total of 229 patients were randomized in this study, but 18 patients were excluded in safety evaluation. Because 17 of them didn't take any study medication (vytorin or atorvastatin) after randomization and one of them couldn't categorize in any group.
Arm/Group | Vytorin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/108 | 5/103
Other Adverse Events (participants affected / at risk) | 19/108 | 22/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vytorin (N=108) | Atorvastatin (N=103)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Thrombosis in device (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vytorin (N=108) | Atorvastatin (N=103)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Infections and infestations) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Generalized oedema (General disorders) | 0 (0) | 2 (2)
Application site reaction (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.